CLINICAL TRIAL: NCT04191889
Title: A Prospective, Single-arm, Phase II Trial to Evaluate the Effectiveness and Safety of Hepatic Arterial Infusion Chemotherapy (HAIC) of Oxaliplatin, 5-fluorouracil and Leucovorin (mFOLFOX7) Combined With Apatinib-Mesylate Tablets and Camrelizumab for Injection for C-staged Hepatocellular Carcinoma in BCLC Classification.
Brief Title: A Trial of Hepatic Arterial Infusion Combined With Apatinib and Camrelizumab for C-staged Hepatocellular Carcinoma in BCLC Classification
Acronym: TRIPLET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yang-kui Gu, Associate Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIPLET
Record Dates: First submitted 2019-12-03; First posted 2019-12-10 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: C-staged Hepatocellular Carcinoma in BCLC Classification
Keywords: Advanced hepatocellular carcinoma; hepatic arterial infusion chemotherapy; anti-PD-1 immunotherapy; Camrelizumab; anti-angiogenic targeted therapy; Apatinib
MeSH Terms: interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRIPLET (Experimental): Hepatic Arterial Infusion combined with Apatinib and Camrelizumab
  Interventions: Combination Product: Hepatic Arterial Infusion combined with Apatinib and Camrelizumab

INTERVENTIONS:
Combination Product: Hepatic Arterial Infusion combined with Apatinib and Camrelizumab — Drug: FOLFOX Protocol (Oxaliplatin, fluorouracil, and leucovorin); Camrelizumab for injection and Apatinib-Mesylate Tablets
  Procedure:
  1. On the first day of treatment, HAIC was conducted through a catheter intubated into the tumor feeding artery under DSA guidance with the following chemotherapeutic drugs (mFOLFOX7, oxaliplatin 85 mg/m2 2 hours, folinic acid 400 mg/m2, 5-FU 2500 mg/m2 46 hours) pumped into the tumor artery. The HAIC is repeated every 3 weeks. The cumulative maximum sessions of HAIC is up to 6 times.
  2. Taking Apatinib-Mesylate Tablets (250 mg/tablet) orally on day 8 in the first HAIC cycle, once a day, for continuous medication.
  3. The first dose of Camrelizumab was administered on day 4 of the second HAIC cycle, at a dose of 200 mg intravenously, every three weeks.
  4. The cumulative maximum drug use period is up to 2 years. The patient is concurrent on medication until the treatment discontinuation criteria specified in the protocol appear.

SUMMARY:
This study was designed to evaluate the effectiveness and safety of hepatic arterial infusion chemotherapy combined with Apatinib and Camrelizumab (Triplet-combined Therapy) for C-staged Hepatocellular Carcinoma in BCLC classification.

The primary outcome measure is to evaluate the objective response rate (ORR) of Triplet-combined Therapy for C-staged Hepatocellular Carcinoma in BCLC classification.

The secondary Outcome measures include the duration of response (DOR), disease control rate (DCR), progression-free survival rate (PFSR) [ Time Frame: 6- and 12-month], overall survival rate (OSR) [ Time Frame: 6- and 12-month], the median progression-free survival time (mPFS) and median overall survival time (mOS) of Triplet-combined Therapy for C-staged Hepatocellular Carcinoma in BCLC classification.

Moreover, this study aims to assess the safety and tolerability of Triplet-combined Therapy for C-staged Hepatocellular Carcinoma in BCLC classification.

DETAILED DESCRIPTION:
Primary liver cancer is a common malignant tumor of the digestive system in the world. There are about 854,000 new incidences and 810,000 mortality each year. In China, there is a high incidence of liver cancer, with about 466,000 new cases and 422,000 mortality each year. Hepatocellular carcinoma (HCC) accounted for about 90% of primary liver cancer in pathological type. Most patients have reached advanced stage or with distant metastasis when diagnosed and the natural median survival time is only 3 to 4 months. Then only systemic therapy is recommended for patients in advanced HCC in many global guidelines.

Hepatic arterial infusion chemotherapy (HAIC) of mFOLFOX7, anti-angiogenic targeting drugs, and antibody immunotherapy against programmed death molecule-1 (PD-1) immunological checkpoints are effective treatment options for advanced hepatocellular carcinoma. Many clinical studies have shown that the two-two combination of the above three treatment options can improve the anti-tumor overall response rate, the survival rate and even achieve clinical complete remission of patients with advanced HCC.

Shi Ming et al reported HAIC combined with systemic targeted therapy has a better survival outcome compared to systemic targeted therapy mono-therapy [OS 13.37 vs 7.13 months, PFS 7.03 vs 2.6 months] in JAMA Oncology. Although the toxicity of combination therapy is slightly higher than that of sorafenib monotherapy, these adverse effects are tolerable.

In addition, in a phase Ib study of Camrelizumab combined with apatinib in the treatment of advanced liver cancer, gastric cancer or gastroesophageal junction cancer showed that in 16 patients with HCC, the ORR was 50.0% and the DCR was 93.8%. When the dose of apatinib was 250 mg, the median PFS was 7.2 months. Camrelizumab combined with low dose apatinib can effectively reduce the incidence of adverse reactions, ≥10% of patients have treatment-related adverse reactions (all levels), no treatment-related adverse reactions leading to death. Therefore, low-dose anti-angiogenic drugs can inhibit tumor angiogenesis on the one hand, reduce immunosuppression by inducing normalization of blood vessels, enhance effector immune cell infiltration, and enhance anti-tumor immunity.

In summary, for patients of C-staged Hepatocellular Carcinoma, HAIC, anti-angiogenic targeted therapy, and anti-PD-1 immunotherapy have their important status, and the combination of any two treatments brings about synergy effect. Then, could the combination of the three treatment methods further improve the outcome of advanced hepatocellular carcinoma? This study was designed to evaluate the efficacy and safety of a combination of hepatic arterial infusion chemotherapy, targeted drugs (Apatinib), and anti-PD-1 immunotherapy (Camrelizumab) to provide a more effective and toxic-tolerable treatment for patients in C-staged Hepatocellular Carcinoma in BCLC classification.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily joins the study and signs an informed consent;
2. Age ≥ 18 years old, ≤ 70 years old, both men and women;
3. Clinical or pathologically confirmed BCLC C-stage hepatocellular carcinoma, no further first-line treatment;
4. At least one intrahepatic evaluable tumor existed, intrahepatic tumor is the primary tumor burden;
5. Child-Pugh score small or equal to 7 points (Child-Pugh A-B);
6. The liver tumor burden does not exceed 50% of the total liver volume;
7. Patient can swallow tablet normally;
8. ECOG score: 0 to 1 (according to the ECOG score classification);
9. The expected survival is longer than 12 weeks;
10. The laboratory parameters meets the following requirements (no blood components and cell growth factors are allowed within 14 days before the first dose):

    * Absolute neutrophil count ≥ 3.0 × 109 / L;
    * Platelets ≥ 80 × 109 / L;
    * Hemoglobin ≥ 90 g / L;
    * serum albumin ≥ 28 g / L;
    * Thyroid stimulating hormone (TSH) ≤ 1 × ULN (if abnormalities should be considered at the same time FT3, FT4 levels, patients with FT3 and FT4 levels in normal range can also be enrolled);
    * bilirubin ≤ 1.5 × ULN (within 7 days prior to the first dose);
    * ALT ≤ 3 x ULN and AST ≤ 3 x ULN (within 7 days prior to the first dose);
    * AKP ≤ 2.5 × ULN; serum creatinine ≤ 1.5 × ULN;
11. For female that non-surgical sterilization or in childbearing age need to use a medically approved contraceptive (such as an intrauterine device, contraceptive or condom) during the study period and within 3 months after the end of the study treatment period; For female that non-surgical sterilization or in childbearing age must have a negative serum or urine HCG test within 72 hours prior to study enrollment; and must be non-lactating; for male patients whose partner in a childbearing age, effective methods of contraception should be given during the trial and at the end of Camrelizumab injection.

Exclusion Criteria:

1. The patient has any active auto-immune disease or a history of auto-immune disease (such as the following, but not limited to: auto-immune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroid hyperfunction; patients with vitiligo. For patient with history of asthma, complete remission of asthma in childhood without any intervention after adulthood can be included, while those asthma patients who require bronchodilators for medical intervention cannot be included.);
2. The patient is using immunosuppressive agents or systemic hormonal therapy for immunosuppression purposes (dose > 10 mg/day of prednisone or other therapeutic hormones) and continues to be used within 2 weeks prior to enrollment;
3. Severe allergic reactions to other monoclonal antibodies;
4. Known for a history of central nervous system metastasis or hepatic encephalopathy;
5. Having a history of organ transplantation;
6. Patients with clinically symptomatic ascites who require puncture, drainage, or ascites drainage within 3 months, except for those who have a small amount of ascites but no clinical symptoms;
7. Suffering from hypertension, and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥90 mmHg);
8. Suffering heart diseases with clinical symptoms or those not well controlled, such as: (1) heart failure in NYHA class 2 or higher; (2) unstable angina; (3) myocardial infarction occurred within 1 year; (4) clinically symptomatic supraventricular or ventricular arrhythmia requiring treatment or intervention; (5) Tc > 450ms (male); QTc > 470ms (female);
9. Coagulation dysfunction (INR>2.0, PT>16s), bleeding tendency or receiving thrombolysis or anticoagulant therapy, allowing prophylactic use of low-dose aspirin or low molecular heparin;
10. There are significant clinically significant bleeding symptoms or clear bleeding tendency within 3 months before enrollment, such as hemoptysis of 2.5ml or more per day, gastrointestinal bleeding, esophageal varices with bleeding risk, hemorrhagic gastric ulcer or vasculitis, etc. If the fecal occult blood is positive in the baseline period, it can be watched, then gastroscope is needed for those fecal occult blood is still positive. If the gastroscope indicates severe esophageal varices, it cannot be enrolled, except for those who have undergone gastroscopy within a month or less to exclude such cases);
11. Events of arterial/venous thrombosis occurring within the first 6 months of enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
12. There are known hereditary or acquired bleeding and thrombophilia (such as hemophilia patients, coagulopathy, thrombocytopenia, etc.);
13. Urine routine indicates that urine protein ≥ ++ and 24-hour urine protein amount > 1.0g was confirmed;
14. The patient has active infection, unexplained fever (≥38.5 °C) within 3 days before administration, or baseline white blood cell count>15×109/L; 15 Patients with congenital or acquired immunodeficiency (such as HIV-infected patients);

16. HBV-DNA>2000 IU/ml (or 104 copies/ml); or HCV-RNA>103 copies/ml; or HBsAg+ and anti-HCV antibody positive patients; 17. The patient has had other malignant tumors in the past 3 years or at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ); 18. Patients with bone metastases who had received palliative radiotherapy >4% of the bone marrow area within 4 weeks prior to participation in the study; 19. Patients have previously received other anti-PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1, or have received apatinib before; 20. Inoculation of a live vaccine within less than 4 weeks prior to study or possibly during the study period; 21. Pregnant or lactating women, or women of childbearing age who are unwilling to take contraceptive measures; 22. According to the investigators, the patient has other factors that may affect the results of the study or lead to the termination of the study, such as alcohol abuse, drug abuse, other serious diseases (including mental illness) requiring combined treatment, and serious laboratory tests, abnormalities, accompanied by factors such as family or society, which may affect the safety of enrolled patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 | From date of first dose of study drug until disease progression (up to approximately 3 years)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1.

SECONDARY OUTCOMES:
Objective response rate (ORR) by mRECIST | From date of first dose of study drug until disease progression (up to approximately 3 years)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by mRECIST.
The disease control rate (DCR) | From date of first dose of study drug until disease progression, stable disease (up to approximately 3 years)
  DCR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1 and mRECIST.
The time to response (TTR) | From date of first dose of study drug to the date of first documentation of CR or PR (up to approximately 3 years)
  TTR was calculated as the time from treatment initiation to first documented response as assessed by RECIST 1.1 and mRECIST.
Duration of response (DOR) by RECIST 1.1 and mRECIST | From the first documentation of CR or PR to the first date of documentation of disease progression or death whichever occurs first (up to approximately 3 years)
  DOR is defined as the time from the first documentation of CR or PR to the date of first documentation of disease progression as assessed by RECIST 1.1 and mRECIST or death (whichever occurs first).
The progression-free survival time (PFS) | From date of first dose of study drug to the date of first documentation of disease progression or death (up to approximately 3 years)
  The progression-free survival time (PFS) defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1 and mRECIST or death, whichever comes earlier.
The liver-specific progression-free survival time (liver-specific PFS) | From date of first dose of study drug to the date of first documentation of disease progression within the liver or death (up to approximately 3 years)
  The liver-specific PFS was defined as the time from treatment initiation to disease progression within the liver as assessed by RECIST 1.1 and mRECIST or death, whichever comes earlier.
The median overall survival time (OS) | From the start date of the Treatment Phase until date of death from any cause (up to approximately 3 years)
  OS is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date.
The progression-free survival rate (PFSR) by RECIST 1.1 and mRECIST | From date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurs first (up to approximately 3 years)
The overall survival rate (OSR) | From date of first dose of study drug to the date of documentation of death from any cause (up to approximately 3 years)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From the start date of the Treatment Phase until date of death from any cause (up to approximately 3 years)
Exploratory outcome measure: The quality of life (QoL) | From date of first dose of study drug to the date of first documentation of disease progression within the liver or death (up to approximately 3 years)
  The exploratory endpoint was the QoL, which was assessed using the European Organisation for Research and Treatment of Cancer QoL questionnaire (EORTC QLQ-C30).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lyu N, Kong Y, Mu L, Lin Y, Li J, Liu Y, Zhang Z, Zheng L, Deng H, Li S, Xie Q, Guo R, Shi M, Xu L, Cai X, Wu P, Zhao M. Hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin vs. sorafenib for advanced hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):60-69. doi: 10.1016/j.jhep.2018.02.008. Epub 2018 Feb 20. PMID 29471013
- [Background] He M, Li Q, Zou R, Shen J, Fang W, Tan G, Zhou Y, Wu X, Xu L, Wei W, Le Y, Zhou Z, Zhao M, Guo Y, Guo R, Chen M, Shi M. Sorafenib Plus Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin vs Sorafenib Alone for Hepatocellular Carcinoma With Portal Vein Invasion: A Randomized Clinical Trial. JAMA Oncol. 2019 Jul 1;5(7):953-960. doi: 10.1001/jamaoncol.2019.0250. PMID 31070690